CLINICAL TRIAL: NCT07060586
Title: The Effect of Sphenopalatine Ganglion Block Versus Placebo on Headache the Day After Participation in Metal Festival: a Randomised Controlled Trial
Brief Title: The Effect of Sphenopalatine Ganglion Block on Headache and Vasalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Christian S. Meyhoff, MD, PhD, Professor, University Hospital Bispebjerg and Frederiksberg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPGCPHHell
Record Dates: First submitted 2025-06-23; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Vasalgia; Headache; Hangover
Keywords: Hangover; SPGB
MeSH Terms: conditions — Headache | interventions — Sphenopalatine Ganglion Block

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Block (Lidocaine + Ropivacaine) (Experimental)
  Interventions: Procedure: Sphenopalatine Ganglion Block
- Sham block (Saline) (Sham Comparator): Incomplete block with saline (no contact with ganglion)
  Interventions: Procedure: Sham Block

INTERVENTIONS:
Procedure: Sphenopalatine Ganglion Block — A bilateral transnasal sphenopalatine ganglion block with cotton tips soaked in a mixture of 0.5 mL lidocaine 4% and 0.5 mL ropivacaine 0.5% plus injection through the cotton tips of an additional 1 mL of the mixture. The Danish Medicines Agency waived need for approval as this procedure is not considered a pharmaceutical intervention.
  Arms: Block (Lidocaine + Ropivacaine)
Procedure: Sham Block — A sham block with two bilaterally inserted cotton tips not reaching the posterior part of the nasopharyngeal making not contact with the ganglion. Cotton tips are soaked in 1 mL placebo (saline) and have a total of 1 mL saline injected through the cotton tips. The Danish Medicines Agency waived need for approval as this procedure is not considered a pharmaceutical intervention.
  Arms: Sham block (Saline)

SUMMARY:
The purpose of this study is to evaluate the effect of sphenopalatine ganglion block (SPG block) on headache and veisalgia (hangover) the day after attending the metal festival Copenhell.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of sphenopalatine ganglion block (SPG block) on headache and veisalgia (hangover) the day after attending the metal festival Copenhell.

Headache is one of the most commonly reported symptoms following heavy alcohol consumption and is expected to be particularly pronounced after exposure to noisy environments. Headaches can have negative consequences such as reduced cognitive function and absence from school or work despite treatment with basic pain medication.

A Danish study has previously shown that SPG block is effective against some of the most severe types of headache (e.g., post-dural puncture headache and migraine), but its potential after participation in a music festival has not yet been explored.

The mechanism and pathophysiology behind headache and veisalgia after significant alcohol intake are not well understood but are believed to be multifactorial. Headache following alcohol consumption is thought to arise from a dysreflexia that leads to cerebral vasodilation, which causes the headache. This cerebral vasodilation is mediated by the parasympathetic nervous system, partly via neurons in the sphenopalatine ganglion (SPG), which is located at the back of the nasal cavity.

Treatment that inhibits this vasodilation by blocking the SPG is still relatively new in Denmark, but a Danish study has demonstrated its effect on post-dural puncture headache, where it was found to potentially cure more than half of the cases, thus sparing patients further invasive treatment. However, the study concluded that much of the block's effect could not necessarily be attributed to the local anesthetic but might instead be due to mechanical stimulation of the ganglion.

In addition to its effect on post-dural puncture headache, the block has also been shown to be effective in migraine, where a similar mechanism is assumed.

The treatment with transnasal sphenopalatine ganglion block (SPG block) is simple and minimally invasive, performed by gently inserting a cotton swab with local anesthetic through the patient's nostril to the back wall of the nasal cavity where the ganglion is located. The block has few reported side effects and can be performed with minimal resources.

ELIGIBILITY:
Screening Criteria:

* Age ≥ 18 years
* Expected to consume a large amount of alcohol at the metal festival Copenhell
* Expected to be able to cooperate during block administration
* No known history of migraine, chronic headache, or allergy to substances used in the study
* Able to understand and speak Danish

Inclusion Criteria:

* Meets screening criteria and is present on the day of intervention
* Moderate to severe headache (defined as ≥ 3 on a 0-10 VAS) on the day of intervention

Exclusion Criteria:

* Intake of alcohol or other intoxicating substances after waking up on the day of intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2025-06-18 (Actual); Primary Completion 2025-06-21 (Actual); Study Completion 2025-06-21 (Actual)

PRIMARY OUTCOMES:
Headache Pain Intensity 10 minutes after SPGB | 10 minutes following block
  Pain intensity (0-100 mm on a visual analog scale, VAS) of the headache in a standing position 10 minutes after administration of the block in the Ropivacaine-Lidocaine group and the Sham group.
  Pain intensity is measured as the worst pain experienced after the person has been standing for 30 seconds, or as the worst pain during the attempt to stand if the test must be aborted.

SECONDARY OUTCOMES:
Pain score below 30mm (VAS) | 10 minutes following block
  Frequency of individuals with a pain score below 30 mm in a standing position (on a visual analog scale, VAS, 0-100 mm ) at 10 minutes after block administration.
Difference in headache pain intensity in standing position | 10 minutes following block
  Difference in pain intensity (0-100 mm on a visual analog scale, VAS) of the headache in the standing position 10 minutes after administration of the block in the Ropivacaine-Lidocaine group and the Sham group. Pain intensity is measured as the worst pain experienced after the person has been standing for 30 seconds, or as the worst pain during the attempt to stand if the test must be aborted. The difference is calculated as the pain intensity after the block minus the pain intensity at baseline before the block.
Severity of veisalgia | 10 minutes following block
  The severity of veisalgia (assessed using the Alcohol Hangover Severity Scale (AHSS)) 10 minutes after block administration. Range of AHSS, 0-120, higher scores worst.
Difference in veisalgia severity | 10 minutes following block
  Difference in vasalgia (assessed using the Alcohol Hangover Severity Scale (AHSS)) 10 minutes after block administration. Range of AHSS, 0-120, higher scores worst.

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhell 2025, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Only if data sharing is accepted by Data Mangement Agency upon request.